CLINICAL TRIAL: NCT06590506
Title: High Definition Medicine: Establishment of a Cohort of Patients With Advanced Cancer for Prospective High-resolution Follow-up
Brief Title: High Definition Medicine for Solid Tumors Oncology
Acronym: HDM-PMP22
Status: Recruiting | Type: Observational
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Responsible Party: Sponsor
Other Study IDs: High Definition Medicine PMP22; PMP22/00032 (Other Grant/Funding Number: Instituto de salud Carlos III)
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Solid Tumor; Advanced Cancer
Keywords: Lung cancer metastatic disease any first line treatment; Colon cancer metastatic disease any first line treatment; Breast cancer luminal first line hormonal treatment + CDK4/6 inhibitor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetics: (tumor biopsy) NGS panel of 52 genes. Circulating nucleotides: (peripheral blood) circulating DNA. Epigenomics: (peripheral blood) changing the DNA sequence. Immunoma: (peripheral blood) level of lymphocytes including B, T, NK and CD45RO lymphocytes and macrophages as well as cytokines (IL-4, IL-5, IL-6, IL-10, IL-13 (anti-inflammatory), IL -2, IL-12 and IFN-ɣ (pro-inflammatory)).
  Metabolome: (peripheral blood) Proteome: (peripheral blood and tumor biopsy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First line breast cancer metastatic subtype luminal: Women with hormone-positive, HER2-negative breast cancer who will receive CDK4/6 inhibitor plus hormone treatment.
  Interventions: Device: Wearable
- First line colon cancer metastatic: Women with colon cancer of any subtype, candidates to receive first-line treatment.
  Interventions: Device: Wearable
- First line lung cancer metastatic: Women with lung cancer of any subtype, candidates to receive first-line treatment.
  Interventions: Device: Wearable

INTERVENTIONS:
Device: Wearable — Continuous monitoring thought data recorded with wearable (Vivosmart Garmin bracelet)
  Other Names: Vivosmart Garmin bracelet

SUMMARY:
The present study aims to analyze different genetic, phenotypic, environmental, social and lifestyle characteristics of cancer patients who are going to start a first line of cancer treatment with palliative intent and their possible relationship with tumor response or tolerance to treatment. In this way, the aim is to identify a series of variables that allow a better selection of patients and oncological treatments.

DETAILED DESCRIPTION:
The objective of this study is to obtain a cohort of patients with advanced cancer that is robust and large enough to study the nature and possible interrelation between these variables and their influence on the response and tolerance to treatment.

To do this, the investigators will rely on the first of the high-definition medicine strategies and evaluate the main health determinants of each individual.

This strategy will be use because by obtaining a personal baseline from a sufficiently large cohort of patients the investigators will be able to interrelate and identify those variables that have greater weight when it comes to obtaining a response or good tolerance to oncological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of oncological disease of solid origin, candidate for first-line treatment (TREATMENT VIRGIN FOR METASTIC DISEASE).
* Advanced tumor stage (III or IV) not a candidate for treatment with curative intent.
* Preference will be given to the following pathologies and sub-types:
* Women with hormone-positive, HER2-negative breast cancer who will receive a CDK4/6 inhibitor plus a hormone inhibitor. o Women with lung cancer of any subtype, candidates to receive first-line treatment.
* Women with colon cancer of any subtype, candidates to receive first-line treatment.
* Patients who are going to start treatment in a clinical trial are allowed, as long as the treatment is known (in other words, patients who participate in double-blind studies would not be candidates). There are no inclusion problems for patients who have different types of therapies within the trial as long as they are known (examples such as the following, but not limited to these: women starting treatment for breast cancer with a SERD and an approved CDK4/6 inhibitor , women who start an AI and an experimental CDK4/6/2, women who start a triplet for breast cancer but include AI+CDK4/6i, women who start a triplet for lung cancer with chemotherapy, pembrolizumab, and an experimental immunotherapy , etc).
* ECOG performance status <2.
* Sufficient capacity and knowledge to carry and use the wearable.
* Have a mobile device with internet access and an email account.
* Ability to complete quality of life, nutrition and mental health questionnaires.
* Written informed consent to participate in the trial obtained prior to any study-specific screening procedures.
* Patients with co-morbidities are not excluded - they are part of the "real world" clinic and it is necessary to know their evolution.
* For the same reason, pregnant women are not excluded.

Exclusion Criteria:

* Having previously received oncological treatment for metastatic disease or with palliative intent.
* Planned participation in treatment in a double-blind trial regime.
* Previous or concomitant malignant disease of any other type that could affect compliance with the protocol or interpretation of results. Patients with curatively treated basal cell carcinoma of the skin or cervical cancer in situ are eligible for the study.
* Concurrent illnesses that may significantly interfere with participation in the study at the discretion of the investigator. No specific diseases are specified, since patients with multiple pathologies are part of the daily clinic and it is very interesting to collect data from patients with other comorbidities, as long as they have the necessary digital familiarization to wear the wearable and use the APP.
* Carriers of therapeutic electronic devices: pacemakers, defibrillators or cardiac resynchronizers (due to potential interference caused by the device).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced incurable and metastatic disease selected with the aim of being able to carry out continuous follow-up from the beginning of the first line of treatment until death or withdrawal of consent; sensing that the duration of follow-up will be acceptable in relation to the life expectancy of these patients.
  Purpose of bringing together a heterogeneous group of tumor stages (locally advanced and metastatic) and tumor origins (breast, colon, lung...) is to obtain data that is sufficiently broad and representative to allow the identification of common risk factors patients of different stages and tumor origins without initially assuming that the origin or stage is a determining factor when tolerating or responding to oncological treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Solid cohort of clinical, analytical and epidemiological variables | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  To generate a large and solid cohort of clinical, analytical and epidemiological variables in patients with advanced cancer breast, lung and colon

SECONDARY OUTCOMES:
Recorded heart rate | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  The feasibility of collecting heart rate using activity bracelets (wareables)
Recorded oxygen saturation | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  The feasibility of collecting oxygen saturation using activity bracelets (wareables)
Recorded physical activity: number daily steps, distance traveled, number steps climbed, and time of physical activity | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  The feasibility of collecting physical activity using activity bracelets (wareables).
  Average time of physical activity: It is the average time, measured in minutes, that the patient remains active. It is a variable that aims to show how long, on average, the individual is capable of maintaining continuous physical activity.
Recorded daily sleep time and quality | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  The feasibility of collecting daily sleep using activity bracelets (wareables). It consists of measuring the hours of daily sleep and the duration of each of the sleep phases. Normal sleep consists of two phases that repeat cyclically: the non-REM (NREM) phase, defined as the non-rapid eye movement phase of sleep; and the REM phase or rapid eye movement sleep phase. Monitoring sleep hours and quality by analyzing vital signs during sleep can detect sleep abnormalities and their correlation with the patient's quality of life.
Adherence to wearable | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  Evaluate the porcentage of patient who meet the adherence to wear wearable monitoring. Measure the time that the patient wears the wearable throughout the study 24 hours a day (with the exception of the times necessary to recharge the battery). The included patients must commit to wearing the wearable for the entire time established in the protocol to optimize their quality and the results obtained.
Correlation Performance Status | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  Correlation between the Performance Status determined by the clinician and the patient's daily activity level.
  The activity tracker will record your step count for each day. The investigators will plot the average daily step count and 95% confidence interval over the entire study period. You will then study the change in step count trajectory during the study. A linear mixed model will be used to describe change over time..
Quality of life questionnaires: EORTC QLQ-C30, Goldberg-GHQ28, Mediterranean diet adherence questionnaire and PRO-CTCAE | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  Correlation between the quality of life reported by the patient through QLQ questionnaires (EORTC QLQ-C30, Goldberg-GHQ28, Mediterranean diet adherence questionnaire and PRO-CTCAE) and the data collected through wearables
Patients' physical routine | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  Identify changes in patients' physical routine throughout the monitoring period: The activity tracker will record your step count for each day. The investigators will plot the average daily step count and 95% confidence interval over the entire study period. You will then study the change in step count trajectory during the study. A linear mixed model will be used to describe change over time.
Correlation of physical activity and tolerance and response to treatment | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  Correlation between the patient's degree of physical activity and tolerance and response to treatment
Correlation of physiological adaptation to exercise and tolerance and response to treatment | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first assessed up to 36 months
  Correlation between the patient's physiological adaptation to exercise and tolerance and response to treatment
Correlation tumor stage and tolerance and response to treatment | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  Correlation between tumor stage and tolerance and response to treatment
Correlation tumor origin and tolerance and response to treatment | From date of inclusion until the date of death from any cause or the date patient withdrawal, whichever came first, assessed up to 36 months
  Correlation between tumor origin and tolerance and response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Quintela, PhD, Principal Investigator — CNIO- Spanish Research Cancer Center
Locations (9):
- Spain (9):
  - Hospital Universitario A Coruña, A Coruña, A Coruña/ Galicia
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Son Espases, Palma de Mallorca, Mallorca / Baleares
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Virgen de la Macarena, Seville, Sevilla/ Andalucia
  - ICO Hospitalet Bellvitge, Barcelona
  - Hospital San Pedro Alcántara de Cáceres, Cáceres
  - Hospital de La Princesa, Madrid
  - Hospital General de Valencia, Valencia